CLINICAL TRIAL: NCT02690649
Title: Keep it SIMPLE: Improving Anti-Coagulation Medication Adherence for Patients With Non-valvular Atrial Fibrillation
Brief Title: Keep it SIMPLE: Improving Anti-Coagulation Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tammy Toscos (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Tammy Toscos, Research Scientist, Informatics, Parkview Health
Organization: Parkview Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRC15-0709
Record Dates: First submitted 2016-02-10; First posted 2016-02-24 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation; Medication Adherence
Keywords: anticoagulants; Personal Health Records
MeSH Terms: conditions — Atrial Fibrillation; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Messaging (Non-Procedural) (Experimental): PHR messaging of tailored health education pertinent to non-valvular atrial fibrillation and anticoagulant use.
  Training on the use of MyChart and the AdhereTech smart pill bottle, medication adherence monitored with Surescripts e-prescribing software and AdhereTech smart pill bottle use.
  Interventions: Other: Health Messaging (Non-Procedural)
- No Health Messaging (No Intervention): No PHR messaging of tailored health education pertinent to non-valvular atrial fibrillation and anticoagulant use.
  Standard care, training on the use of MyChart and the AdhereTech smart pill bottle, medication adherence monitored with Surescripts e-prescribing software and AdhereTech smart pill bottle use

INTERVENTIONS:
Other: Health Messaging (Non-Procedural) — Tailored health messaging delivered via the PHR MyChart pertinent to non-valvular atrial fibrillation and anticoagulant use. Messages will be triggered by medication non-adherence information obtained from Surescripts e-prescribing data and use of AdhereTech smart pill bottle.
  Arms: Health Messaging (Non-Procedural)

SUMMARY:
This is an interventional study designed to develop patient focused strategies that improve adherence to anticoagulant medication in patients with non-valvular atrial fibrillation (AF). Outcomes of this work include a novel intervention, as well as information regarding patient preferences for tailored education.

DETAILED DESCRIPTION:
This is an interventional study designed to develop patient focused strategies that improve adherence to anticoagulant medication in patients with non-valvular atrial fibrillation (AF). Outcomes of this work include a novel intervention, as well as information regarding patient preferences for tailored education.

There will be two phases in this study. In the first phase, the investigators will use a patient-centered approach to design and build a personal health record (PHR)-based educational intervention based on patient preferences for content, timing and delivery mechanism. In the second phase, the investigators will test the intervention in a six-month randomized controlled trial.

During the development of the intervention in Phase 1 the investigators will use a patient-centered, iterative design process that includes interviews, prototype development and testing. The investigators will recruit a diverse group of AF patients to determine preferences for information about AF and anticoagulant therapy. The investigators will use a user-centered design approach and best practices in human-computer interactions (HCI) to determine the desired content, timing, and delivery of tailored education in the PHR. The investigators will build out wire-frame models (low fidelity messaging prototypes) based on focus group findings to perform usability testing and further refine the intervention design. The intervention component will assess the impact of pushing tailored health education messages to patients through their PHR. The tailored health education will be specifically aimed at improving patient compliance with anticoagulant therapy.

One trigger for health education messaging will be failure to take, fill, or refill anticoagulant medication prescription - information obtained from an e-prescribing data feed to the electronic medical record (Surescripts) and use of a smart pill bottle (AdhereTech - HIPAA compliant, FDA-registered Class I medical device) that sends notification in real time when participants open or fail to open their pill bottle.

The intervention trial in Phase 2 will be comprised of two groups, control and experimental. Both the control and experimental group will receive standard care, which includes access to MyChart. In addition to standard care, both groups will receive training on the use of MyChart and the AdhereTech smart pill bottle, and medication adherence for both groups will be monitored with Surescripts e-prescribing software and AdhereTech smart pill bottle use. The experimental group will receive the intervention: tailored health messaging delivered via MyChart pertinent to AF and oral anticoagulant use.

ELIGIBILITY:
FOCUS GROUPS:

Inclusion Criteria:

1. Diagnosis of Atrial Fibrillation (Paroxysmal, Persistent, Permanent)

   * focus groups 1 & 2: patients diagnosed ≤ 6 months
   * focus groups 3 & 4: patients diagnosed ≥ 6 months
2. Receiving Oral Anticoagulation -Vitamin K Antagonist (VKA) or Novel Oral Anticoagulant (NOAC)- for non-valvular AF

   * focus groups 1 & 2: on VKA or NOAC
   * focus groups 3 & 4: changed VKA to NOAC within last 6 months
3. *Physically and Mentally capable of providing Informed Consent
4. *Age 18 years or older
5. *Ability to read and understand English
6. Current Patient of Parkview Physicians Group (PPG)-Cardiology

   * 3, 4, and 5 must apply to caregivers, partners, and/or support persons

Exclusion Criteria:

1. Absence of History of Atrial Fibrillation (AF)
2. *Does not meet Inclusion Criteria
3. Anticoagulation with VKA or NOAC for reasons other than non-valvular AF
4. *Designated as part of a vulnerable subject population that the investigator or designee identifies to have compromised autonomy related to potential study participation
5. Currently participating in another Parkview study that involves PHR use

   * Only 2 and 4 apply to caregivers, partners, and/or support persons

TECHNOLOGY TRIAL:

Inclusion Criteria:

1. Diagnosis of Atrial Fibrillation (Paroxysmal, Persistent, Permanent)
2. Receiving Oral Anticoagulation (VKA or NOAC) for non-valvular AF
3. Physically and Mentally capable of providing Informed Consent
4. Age 18 years or older
5. Access to Computer and Internet
6. Ability to read and understand English
7. Current Patient of PPG-Cardiology
8. Willing to have a MyChart account

Exclusion Criteria:

1. Absence of History of Atrial Fibrillation (AF)
2. Does not meet Inclusion Criteria
3. Anticoagulation with VKA or NOAC for reasons other than non-valvular AF
4. Unable to physically or cognitively carry out the tasks necessary for utilizing a PHR such as; blindness, loss of function of arms, cognitive impairments (per chart review) that would interfere in learning a new task
5. Designated as part of a vulnerable subject population that the investigator or designee identifies to have compromised autonomy related to potential study participation
6. Currently participating in another Parkview study that involves PHR use
7. Not willing to have a MyChart account

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Toscos, PhD, Principal Investigator — Parkview Research Center; Parkview Health; Michael Mirro, MD, Principal Investigator — Parkview Research Center; Parkview Health
Locations (1):
- Parkview Research Center; Parkview Health, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Messaging (Non-Procedural): PHR messaging of tailored health education pertinent to non-valvular atrial fibrillation and anticoagulant use.
  Health Messaging (Non-Procedural): Tailored health messaging delivered via the PHR MyChart pertinent to non-valvular atrial fibrillation and anticoagulant use. Messages will be triggered by medication non-adherence information obtained from Surescripts e-prescribing data and use of AdhereTech smart pill bottle.
- No Health Messaging: No PHR messaging of tailored health education pertinent to non-valvular atrial fibrillation and anticoagulant use.
Period: Overall Study
Arm/Group | Health Messaging (Non-Procedural) | No Health Messaging
Started | 80 | 80
Completed | 79 | 76
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Messaging (Non-Procedural) | No Health Messaging | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.78 (8.65) | 71.51 (8.21) | 71.14 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 49 | 51 | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Atrial Fibrillation Knowledge [Mean (Standard Deviation); unit: units on a scale] — 0 is no knowledge, 11 is high knowledge
  units on a scale | 6.94 (1.93) | 6.59 (2.13) | 6.76 (2.04)
Pre-intervention Patient Portal Logins [Mean (Standard Deviation); unit: logins] | 17.80 (18.83) | 18.60 (20.85) | 18.20 (19.80)
Medication Type [Count of Participants; unit: Participants]
  Warfarin | 40 | 40 | 80
  Xarelto | 17 | 12 | 29
  Eliquis | 23 | 28 | 51
Atrial fibrillation diagnosis in previous 12 months [Count of Participants; unit: Participants]
  Yes | 17 | 7 | 24
  No | 63 | 73 | 136

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: AdhereTech smart pill bottles used to collect medication dosing = percentage of allotted doses that were recorded as taken
Time Frame: 6 months during study
Measure: Mean (Standard Deviation); unit: percentage of doses recorded as taken
Arm/Group | Health Messaging (Non-Procedural) | No Health Messaging
Number analyzed (Participants) | 79 | 76
percentage of doses recorded as taken | 93.08 (0.01) | 89.52 (0.01)
Statistical Analysis 1: Comparison: Health Messaging (Non-Procedural); estimated adherence rate for the intervention group Generalized linear models were used to test the effect of the intervention on medication adherence. These generalized linear models used a Poisson distribution to estimate the rate of adherence with the log of total prescribed doses as an offset term in the linear predictor; Test type: Superiority; p = 0.28, Regression, Linear; estimated adherence rate for the interve = 94, 95% CI 2-sided [92 to 95]

2. Secondary Outcome: Patient Portal Login
Description: The number of times participants logged into their patient portal (Epic's MyChart) during the study period was used as a proxy for patient engagement.
Time Frame: 6 months during study
Measure: Mean (Standard Deviation); unit: Count of MyChart patient portal logins
Arm/Group | Health Messaging (Non-Procedural) | No Health Messaging
Number analyzed (Participants) | 80 | 80
Count of MyChart patient portal logins | 42.7 (37.0) | 15.9 (16.0)
Statistical Analysis 1: Comparison: Health Messaging (Non-Procedural) vs No Health Messaging; Test type: Superiority; p < 0.001, Regression, Linear — A negative binomial distribution because the outcome was a count variable and it was over-dispersed; Age, previous patient portal logins, and gender were used as co-variates in the model

3. Secondary Outcome: Atrial Fibrillation Knowledge
Description: End of study score on Atrial Fibrillation Knowledge scale (min:0 is no knowledge, max: 11 is high knowledge), adjusted for age, baseline knowledge, gender and education level.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Health Messaging (Non-Procedural): PHR messaging of tailored health education pertinent to non-valvular atrial fibrillation and anticoagulant use.
  Training on the use of MyChart and the AdhereTech smart pill bottle, medication adherence monitored with Surescripts e-prescribing software and AdhereTech smart pill bottle use.
  Health Messaging (Non-Procedural): Tailored health messaging delivered via the PHR MyChart pertinent to non-valvular atrial fibrillation and anticoagulant use. Messages will be triggered by medication non-adherence information obtained from Surescripts e-prescribing data and use of AdhereTech smart pill bottle.
Arm/Group | Health Messaging (Non-Procedural) | No Health Messaging
Number analyzed (Participants) | 77 | 72
score on a scale | 7.31 (1.92) | 6.64 (2.00)
Statistical Analysis 1: Comparison: Health Messaging (Non-Procedural) vs No Health Messaging; Test type: Superiority; p = 0.03, Regression, Linear — baseline AF knowledge, gender, age, and educational level were all used as co-variates; generalized linear model tested whether AF knowledge at study completion was related to baseline AF knowledge, gender, age, and educational level; Slope = -0.61, 95% CI 2-sided [-1.14 to -0.07]

4. Secondary Outcome: Number of Patients With Incidence of Adverse Events
Description: Adverse events include death, stroke, any embolic event, and/or major bleeding.
Time Frame: 6 months during study
Measure: Count of Participants; unit: Participants
Arm/Group | Health Messaging (Non-Procedural) | No Health Messaging
Number analyzed (Participants) | 80 | 80
Participants | 11 | 6

ADVERSE EVENTS:
Time Frame: 6 months time of study
Description: The intervention was education only; not clinical.
Arm/Group | Health Messaging (Non-Procedural) | No Health Messaging
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 4/80 | 3/80
Other Adverse Events (participants affected / at risk) | 7/80 | 3/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Messaging (Non-Procedural) (N=80) | No Health Messaging (N=80)
Influenza A (Infections and infestations) | 1 (1) | 0 (0) — Influenza A Hospitalization
GI Bleed (Gastrointestinal disorders) | 2 (2) | 1 (1) — GI Bleed Hospitalization
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) — UTI Hospitalization
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) — Chest Pain Hospitalization
Vascular Parkinsonism with dementia (Nervous system disorders) | 0 (0) | 1 (1) — Vascular Parkinsonism with dementia Hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Messaging (Non-Procedural) (N=80) | No Health Messaging (N=80)
Worsening Dyspnea (Cardiac disorders) | 1 (1) | 0 (0) — Worsening Dyspnea Emergency Room Visit
Vestibular Schwannoma (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Vestibular Schwannoma Emergency Room Visit
Ankle pain, arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Ankle pain, arthritis Emergency Room Visit
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) — Palpitations Emergency Room Visit
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Abdominal pain Emergency Room Visit
Penile and Scrotal Rash (General disorders) | 0 (0) | 1 (1) — Penile and Scrotal Rash Emergency Room Visit
Hematuria (General disorders) | 1 (1) | 0 (0) — Hematuria Emergency Room Visit
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) — Chest Pain Emergency Room Visit
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Atrial Fibrillation Emergency Room Visit
Gout (General disorders) | 1 (1) | 0 (0) — Gout Emergency Room Visit
Diabetes Type 2 (Endocrine disorders) | 0 (0) | 1 (1) — Emergency Room Visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT02690649/Prot_000.pdf